CLINICAL TRIAL: NCT04295694
Title: Effect of Infant Immunization on Procalcitonin Levels
Brief Title: Effect of Infant Immunization on Procalcitonin Levels - A Pilot Study
Status: Completed | Type: Observational
Sponsor: CAMC Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 1997459
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Immunization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Fever is a well-known side effect of immunizations. When a febrile infant presents to a healthcare site, such as an emergency room, a large number of tests are usually performed, which may include a procalcitonin (PCT) level. PCT is being increasingly recognized as an inflammatory marker suggestive of serious bacterial infection, and is being used in clinical practice in the workup for acute febrile illness. Based on an elevated PCT level, further testing may be done, antibiotics may be started, and the patient may get admitted to the hospital for observation before identifying the cause of the elevated PCT level. The investigators believe that immunizations can cause an increase in PCT levels in the absence of an acute infection. Thus, a finding of elevated procalcitonin in a recently immunized child may not have the same clinical implication as it does in other clinical scenarios. To investigate this, the investigators designed this pilot prospective study to compare PCT levels immediately before and forty-eight hours after the administration of routine infant immunizations. The investigators will enroll healthy infants presenting for their two, four, and six-month well child visits at FamilyCare - Children's Medicine Center and receiving routine immunizations as recommended by the Centers for Disease Control.

DETAILED DESCRIPTION:
This pilot study is a prospective study enrolling infants who are currently healthy, have no acute illness in preceding fourteen days, and were born full term that are presenting at FamilyCare - Children's Medicine Center (CMC) for their 2, 4, and 6-month well child visit that includes routine immunizations. Following informed consent, a blood sample will be obtained from enrolled infants for PCT testing prior to their routine, scheduled immunizations. The infants will return to CMC to have their PCT levels re-tested at 2 days post immunization. An infant will be included in the study for only one well child visit; if an infant presents for a subsequent well child visit falling within our sample visit age, the infant is not eligible for study re-enrollment. The parent/guardian will be contacted via telephone at week post second blood draw to determine if the infant has experienced symptoms or received medical care during that time period. The patient population targeted for this pilot study will be infants presenting to their pediatricians at FamilyCare - Children's Medicine Center for two, four, or six-month well child visits on a Monday, Tuesday, or Wednesday and receiving their vaccines as recommended by the 2014 CDC schedule.10 This is a pilot study, and therefore had no power analysis performed to calculate sample size. The investigators anticipate that there will be a high rate of patients not returning for the second blood draw, approximately 50%, based on prior patient experience of the investigators. To achieve the sample of at least 20 patients completing both blood draws and the phone interview, the investigators will enroll 45 patients.

ELIGIBILITY:
Inclusion Criteria:

* • Infants receiving their 2,4, or 6 month well-child visit at FamilyCare-Children's Medicine Center that will include their normal, routine 2, 4, or 6 month immunizations (Prevnar®, Pediarix®, ActiHIB®, Rotateq®)

  * Infant age 8 to 28 weeks old at time of study enrollment
  * infant, with no acute illness (cough, congestion, fever, or decreased oral intake, …etc) in preceding fourteen days
  * Infants born full term (37 weeks or more gestation)

Exclusion Criteria:

* • Infants born premature (born prior to 37th week of gestation)

  * Having symptoms of illness in proceeding fourteen days (cough, congestion, fever, or decreased oral intake, …etc)
  * Any previous hospitalizations, with exception of the hospitalization at birth
  * Sick contacts in the home (contacts with symptoms of cough, congestion, or fever)
  * Infants who received vaccines that are different from the standard vaccines that are administered in Children's Medicine Center, to maintain consistency of the study sample
  * Infants with a chronic illness that increases their risk of infections (bronchopulmonary dysplasia, congenital heart disease, immunodeficiency…)

Ages: 8 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The patient population targeted for this pilot study will be infants presenting to their pediatricians at FamilyCare - Children's Medicine Center for two, four, or six-month well child visits on a Monday, Tuesday, or Wednesday and receiving their vaccines as recommended by the 2014 CDC schedule.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2014-08; Primary Completion 2016-07-01 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
To compare change in PCT levels before and after routine immunization in healthy infants two to six months of age. | 2 months up to 6 months
  a blood sample will be obtained from enrolled infants for PCT testing prior to their routine, scheduled immunizations. The infants will return to CMC to have their PCT levels re-tested at 2 days post immunization.

CONTACTS AND LOCATIONS:
Locations (1):
- FamilyCare HealthCenter Children's Medicine Center, Charleston, West Virginia, United States